CLINICAL TRIAL: NCT01299844
Title: Impact of Type 2 Diabetes Peer Counseling on Behavioral, Metabolic, and Health Outcomes Among Latinos
Acronym: DIALBEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Hartford Hospital (Other); Hispanic Health Council, Inc. (Other)
Responsible Party: Rafael Pérez-Escamilla, Ph.D., Director, Center for Eliminating Health Disparities among Latinos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H05-351
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention)
- Diabetes Peer Counseling (Experimental)
  Interventions: Behavioral: Diabetes Peer Counseling

INTERVENTIONS:
Behavioral: Diabetes Peer Counseling — 16 Home visits from a bilingual/bicultural diabetes peer counselor.
  Other Names: DIALBEST
  Arms: Diabetes Peer Counseling

SUMMARY:
The objectives of this study are:

* To develop a comprehensive culturally tailored model of diabetes management that integrates the work of community-based peer counselors and clinical specialists into a multi-disciplinary health care team serving the Latino community.
* To implement an intervention that provides education and support to Latino adults diagnosed with Type 2 diabetes in both clinical and home settings.
* To evaluate this intervention for its impact on program adherence, and improved outcomes sustained over time as reflected by metabolic, clinical, cognitive and behavioral measures.

DETAILED DESCRIPTION:
A randomized two group longitudinal design with clinical measurements and behavioral assessments collected at baseline, 3,6,12 and 18 months will be used. It is hypothesized that participants in the home-based peer-counseling intervention will have greater reductions and will better maintain their reductions in their HbA1c levels compared to participants in the standard of care hospital based program currently in place. Additional secondary hypotheses state the participants in the home-based peer-counseling intervention will have improved lipid profile values, cholesterol levels, and BMI compared to participants in the standard of care hospital based program.

Participants in the home-based peer-counseling intervention will monitor their glucose more regularly (defined by the mean and variance in number of monitored days per month) than participants in the standard of care hospital based program. Lastly, participants in the home-based peer-counseling intervention will have a higher rate of program participation (defined by adherence to appointments and referrals) and completion than participants in the standard of care hospital based program.

ELIGIBILITY:
Inclusion Criteria:

* Latinos older than 21
* Diagnosed with type 2 diabetes
* Referred to the "Amigos en Salud" program at Hartford Hospital
* Residents of Hartford

Exclusion Criteria:

* Advanced renal failure
* Advanced heart disease
* Diagnosis of major psychological disorder or mental condition
* Limb amputation(s) that prevent following study's exercise recommendations
* Any other health condition that prevents individual from consuming all their meals orally

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Change in Baseline in HbA1c at 6 Months

SECONDARY OUTCOMES:
Diabetes Knowledge Test Score | Change from Baseline in Diabetes Knowledge Test Score at 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pérez-Escamilla, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Perez-Escamilla R, Damio G, Chhabra J, Fernandez ML, Segura-Perez S, Vega-Lopez S, Kollannor-Samuel G, Calle M, Shebl FM, D'Agostino D. Impact of a community health workers-led structured program on blood glucose control among latinos with type 2 diabetes: the DIALBEST trial. Diabetes Care. 2015 Feb;38(2):197-205. doi: 10.2337/dc14-0327. Epub 2014 Aug 14. PMID 25125508